CLINICAL TRIAL: NCT01669317
Title: Mechanisms Underlying the Sleep Promoting Effect of Cherry Juice Standardized to Its Proanthocyanidin Content
Acronym: CHERRY JUICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Cherry Grower's Association (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 12004
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Insomnia; Sleep Problem
Keywords: Cherry Juice Pilot
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cherry Juice Standardized (Experimental): You will be given an 8-ounce glass of cherry juice to drink when you arrive at the Sleep Laboratory.
  Interventions: Other: 8-ounce glass of cherry juice; Other: Artificial Cherry Juice
- Artificial Cherry Juice (Placebo Comparator): You will be given an 8-ounce glass of artificial cherry juice to drink when you arrive at the Sleep Laboratory.
  Interventions: Other: 8-ounce glass of cherry juice; Other: Artificial Cherry Juice

INTERVENTIONS:
Other: 8-ounce glass of cherry juice — You will be given an 8-ounce glass of cherry juice or artificial cherry juice to drink when you arrive at the Sleep Laboratory.
Other: Artificial Cherry Juice — You will be given an 8-ounce glass of artificial cherry juice

SUMMARY:
This study is designed to demonstrate that cherry juice is effective in treating insomnia, and to show that it works by inhibiting an enzyme that will be measured in the blood.

DETAILED DESCRIPTION:
This study will consist of 4 visits - 1 screening visit and 3 treatment visits. Screening visit will consist of a fasting chemistry panel, a health questionnaire, an Insomnia Severity Index, the Epworth Sleepiness Scale, the Pittsburgh Sleep Quality Index, the Beck Depression Inventory, the State-Trait Anxiety Inventory, and the Fatigue Severity Scale.

Ten subjects passing screening will take for 2 weeks between dinner and bedtime in a blinded and balanced order: 1. Eight ounces of cherry juice standardized to its proanthocyanidin content in the morning and 8 ounces of cherry juice standardized to its procyanidin content 1-2 hours before bedtime for 14 days; 2. A similar amount of placebo juice with the same timing for the cross-over. There will be a 2-week washout between each of the treatment periods. Subjects will be scheduled for two overnight PSGs, one at the end of each two-week treatment period. On the morning following each test the insomnia severity index and other questionnaires will be repeated. The order of the placebo juice and cherry juice will be random and balanced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female with a usual bedtime between 9 pm and midnight.
* 65 years of age or older.
* Sleep problem >3 nights per week, meeting the International Classification of Sleep Disorders (ICSD-2*) diagnostic criteria of insomnia for at least 6 months.
* An insomnia severity index ≥ 10 and a minimum of 30 minutes of either sleep-onset latency (SL) or wake after sleep onset (WASO).

  *ICSD-2 general criteria for insomnia:
* A complaint of difficulty initiating sleep, difficulty maintaining sleep, or waking up too early, or sleep that is chronically non-restorative or poor in quality.
* The above sleep difficulty occurs despite adequate opportunity and circumstances for sleep.
* At least one of the following forms of daytime impairment related to the nighttime sleep difficulty is reported by the patient:
* Fatigue or malaise.
* Attention, concentration, or memory impairment.
* Social or vocational dysfunction or poor school performance.
* Mood disturbance or irritability.
* Daytime sleepiness.
* Motivation, energy, or initiative reduction.
* Proneness for errors or accidents at work or while driving.
* Tension, headaches, or gastrointestinal symptoms in response to sleep loss.
* Concerns or worries about sleep.

Exclusion Criteria:

* Diabetes.
* Sedating or hypnotic medications.
* Any chronic medication that has not had a stable dose for 1 month or longer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compare the polysomnography of participants with insomnia | Baseline and Week 4
  Compare the polysomnography of participants with insomnia on a night at the end of 2 weeks taking: Eight ounces of standardized cherry juice vs. the night taking the placebo juice.

SECONDARY OUTCOMES:
Compare the Insomnia Severity Index and validated questionnaires | Baseline and Week 4
  Compare the Insomnia Severity Index, a validated questionnaire, in participants with insomnia on a night at the end of 2 weeks taking: 1. Eight ounces of cherry juice standardized to its proanthocyanidin content in the morning, and 1-2 hours before bedtime; 2. Eight ounces of an identical appearing placebo in the morning and 1-2 hours before bedtime.
Comparison of insomnia sleep scales | Baseline and Week 4
  Compare five different sleep quality scales with insomnia on a night at the end of 2 weeks taking: 1. An 8-ounce glass of cherry juice standardized to its proanthocyanidin content in the morning and 1-2 hours before bedtime; 2. an 8- ounce glass of an identical appearing placebo in the morning and 1-2 hours before bedtime.
Differences in the enzyme blood test | Baseline, Week 2 & Week 4
  compare the expression of enzyme blood test of participants taking the standardized cherry juice vs. the the placebo juice.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States